CLINICAL TRIAL: NCT05065606
Title: Descriptive Analysis of Soft-tissue Urate Deposits, and Bone and Joint Destruction in Dual-energy Computed Tomography Exams of Adult Patients With Gout
Brief Title: Descriptive Analysis of Dual-energy Computed Tomography Exams of Adult Patients With Gout
Acronym: DECTGOUT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP180476
Record Dates: First submitted 2020-11-19; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual-energy computed tomography — Dual-energy scanner examinations stored in the PACS (medical imagery) at Lariboisière Hospital are to be analyzed retrospectively and prospectively

SUMMARY:
The main objective is to describe urate deposits (especially in terms of distribution and volume) in soft tissues and bone, and joint erosions and destruction, in adult patients with gout.

DETAILED DESCRIPTION:
Gout is the result of hyperuricemia, itself a consequence of a disorder of purine metabolism. This hypuricemia can lead to the deposition of sodium urate crystals in the soft tissues. It is the deposition of sodium urate crystals in and near the joints that causes an intense local inflammatory reaction with episodes of acute joint pain, swelling and functional disability. In the long term, uratic concretions in the soft tissues (tophus) occur, the joints are destroyed (uratic arthropathies), the kidneys also (gouty nephropathy).

Dual-energy CT (Computed Tomography) is a relatively recent technique that allows the identification of certain materials through the analysis of the difference in attenuation of the material exposed to two different X-ray spectra. This technique identifies the crystalline component of tophus.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old;
* Patient with a gout according to ACR (American College of Rheumatology) criteria;
* Affiliated with a social security scheme.
* Dual-energy scanner examinations stored in the PACS at Lariboisière Hospital

Exclusion Criteria:

* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of dual-energy CT exams performed in routine care in patients with gout according to ACR criteria, patients included between end of year 2016 and end of year 2021 (retrospective and prospective inclusion, retrospective analysis)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Soft tissue tophus description | The day of the CT (computed tomography) examination
  Description of soft tissue tophus in terms of location, size, density at high and low energy
Distribution of urate deposits | The day of the CT examination
  Distribution of urate deposits in soft tissues and bone, and joint erosions and destruction
Descriptive analysis of joint erosions and destruction | The day of the CT examination
  Descrition of joint erosions and destruction :erosion size (mm) and location (joint), joint destruction (space narrowing, joint collapse, joint ankylosis).

SECONDARY OUTCOMES:
Correlation of the descriptive parameters on dual-energy CT with clinical data | The day of the CT examination
  to correlate the descriptive parameters on dual-energy CT with clinical data, including disease history and therapeutic management, and serum urate level.
Variations in tophaceous burden | The day of the CT examination
  To study the variations in tophaceous burden according to the choice of technical parameters for deposit analysis.The parameters of dual energy analysis (threshold, optional filter to remove noise, gradients of dual-energy) change the quantitative value provided by the manufacturer. This outcome will be the urate volume obtained at different parameters
Link between tophus and erosions | The day of the CT examination
  To analyze the relationships between bone erosion scores and urate volume (correlation between quantitative values)
Reproducibility of a scoring system | The day of the CT examination
  To develop and evaluate the reproducibility of a scoring system for tophaceous load and structural damage using a dual energy CT. We will try to developp a scoring system combining the tophus load (total tophus volume) and the erosion score (total erosion score).
Bone mineral density | The day of the CT examination
  To evaluate the bone mineral density at the distal radius and correlate it with tophaceous load and joint structural damage. A region of interest at the distal radius (one centimeter above the joint space) will be placed using the computer mouse to obtained the bone mineral density (in Hounshield unit, mean bone mineral density within the ROI (Region Of Interest)).
Tophus texture | The day of the CT examination
  To evaluate tophus texture. The texture of the tophus will be approached qualitatively (homogeneous/heterogeneous) and according to its density (Hounsfield unit) and to the percentage of tophus color-coded by the dual energy analyse.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BOUSSON, PUPH, Study Director — APHP Lariboisière - Imagerie OstéoArticulaire,Viscérale; Valérie BOUSSON, PUPH, Principal Investigator — APHP Lariboisière - Imagerie OstéoArticulaire,Viscérale
Locations (3):
- France (3):
  - Hôpital Lariboisière - Service d'Imagerie OstéoArticulaire, Viscérale et Vasculaire, Paris
  - Hôpital Lariboisière - Service de Rhumatologie, Paris
  - Hôpital Bichat - Service de Rhumatologie, Paris

IPD SHARING:
Plan to Share IPD: No